CLINICAL TRIAL: NCT02684981
Title: Non-interventional Study Describing Patients´ Perception on Anticoagulant Treatment and Treatment Convenience When Treated With Pradaxa or Vitamine K Antagonist for Stroke Prevention in Non-Valvular Atrial Fibrillation
Brief Title: Patient Convenience Study (RE-SONANCE)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.249
Record Dates: First submitted 2015-11-11; First posted 2016-02-18 (Estimated); Results first posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-05

CONDITIONS: Atrial Fibrillation; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Cohort A - VKA to Pradaxa switcher: Patients with non-valvular atrial fibrillation (NVAF), currently on Vitamin K Antagonist (VKA) therapy, who are switched to Pradaxa.
- Cohort B - newly assigned to treatment: Newly diagnosed NVAF patients who are treated with VKA or Pradaxa (VKA : Pradaxa = 1:1).

SUMMARY:
The aim of this non-interventional study is to describe patient's perception of anticoagulant treatment when using Pradaxa to prevent stroke and systemic embolism while suffering from atrial fibrillation (according to its approved indication in the approved dosages of 110 milligrams or 150 milligrams twice daily) in comparison to standard care using Vitamin K Antagonist (VKA).

ELIGIBILITY:
Inclusion criteria:

Cohort A:

1. A. Written informed consent prior to participation
2. A. Female and male patients >= 18 years of age with a diagnosis of non-valvular atrial fibrillation.
3. A. At least 3 months of continuous VKA treatment for stroke prevention prior to baseline assessment.
4. A. Patients switched to Pradaxa according Summary of Product Characteristics and physician's discretion.

OR

Cohort B:

1. B. Written informed consent prior to participation.
2. B. Female and male patients >= 18 years of age newly diagnosed with non-valvular atrial fibrillation and no previous treatment for stroke prevention (no use of any oral anticoagulant (OAC) within one year prior to enrolment).
3. B. Stroke prevention treatment initiated with Pradaxa or VKA according to Summary of Product Characteristics and physician's discretion.

Exclusion criteria:

1. Contraindication to the use of Pradaxa or VKA as described in the Summary of Product Characteristics (SmPC).
2. Patients receiving Pradaxa or VKA for any other condition than stroke prevention in atrial fibrillation.
3. Current participation in any clinical trial of a drug or device.
4. Current participation in an European registry on the use of oral anticoagulation in AF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: European patients with non valvular atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 9472 (Actual)
Dates: Start 2015-11-11 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (12):
- Multiple Locations, Austria
- Multiple Locations, Bulgaria
- Multiple Locations, Czechia
- Multiple Locations, Estonia
- Multiple Locations, Hungary
- Multiple Locations, Israel
- Multiple Locations, Latvia
- Multiple Locations, Poland
- Multiple Locations, Romania
- Multiple Locations, Russia
- Multiple Locations, Serbia
- Multiple Locations, Slovenia

REFERENCES:
- [Derived] Vinereanu D, Napalkov D, Bergler-Klein J, Benczur B, Ciernik M, Gotcheva N, Medvedchikov A, Poder P, Simic D, Skride A, Tang W, Trusz-Gluza M, Vesely J. Patient perceptions of anticoagulant treatment with dabigatran or a vitamin K antagonist for stroke prevention in atrial fibrillation according to region and age: an exploratory analysis from the RE-SONANCE study. J Thromb Thrombolysis. 2021 Nov;52(4):1195-1206. doi: 10.1007/s11239-021-02450-2. Epub 2021 Apr 30. PMID 33929686

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an observational study. Total 9472 patients with Non-Valvular Atrial Fibrillation (NVAF) were enrolled in the study using Vitamin K antagonist (VKA) therapy prior to being switched to Pradaxa® and newly diagnosed with NVAF and initiated Pradaxa® or VKA. Patients were followed up for observational period of approximately 6 months.
Pre-assignment Details: All patients were screened for eligibility. All enrolled patients met all implemented inclusion/exclusion criteria. Out of 9472 enrolled patients, 7 patients with unknown study treatment were not included in the main analysis set. Total 9465 patients were included in the main analysis set and started the study.
Groups:
- Cohort A: Patients with Non-Valvular Atrial Fibrillation (NVAF) using Vitamin K Antagonist (VKA) therapy prior to being switched to oral dose of Pradaxa® 110 milligram (mg) and Pradaxa® 150 mg hard capsules twice daily containing Dabigatran etexilate (active ingredient: Dabigatran) were included.
- Cohort B- Pradaxa®: Newly diagnosed patients with Non-Valvular Atrial Fibrillation (NVAF) and initiated Pradaxa® 110 mg and Pradaxa® 150 mg hard capsules twice daily containing Dabigatran etexilate (active ingredient: Dabigatran) therapy.
- Cohort B- VKA: Newly diagnosed patients with Non-Valvular Atrial Fibrillation (NVAF) and initiated Vitamin K Antagonist (VKA) therapy were included.
Period: Overall Study
Arm/Group | Cohort A | Cohort B- Pradaxa® | Cohort B- VKA
Started (Number of patients started are treated with known treatment.) | 4100 | 3179 | 2186
Completed | 3860 | 2969 | 2059
Not Completed | 240 | 210 | 127
Not completed — Permanently discontinued the treatment | 157 | 161 | 110
Not completed — Other | 83 | 49 | 17

BASELINE CHARACTERISTICS:
Population: Main Analysis set (MAS): This includes all eligible patients who met inclusion/exclusion crteria with known assigned treatment information.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B- Pradaxa® | Cohort B- VKA | Total
Number analyzed (Participants) | 4100 | 3179 | 2186 | 9465
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.5 (9.57) | 68.6 (10.1) | 68.5 (9.49) | 69.4 (9.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1998 | 1602 | 1080 | 4680
  Male | 2102 | 1577 | 1106 | 4785
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Convenience PACT-Q2 Scores at Second and Last Assessment Compared to Baseline Assessment
Description: The individual questions in PACT-Q2 were grouped into two domains, convenience and satisfaction. For each domain, a global score was calculated and used for analysis. The range of the global score is 0-100, with higher score indicating better outcome. The global score is calculated by summing up the individual scores, and then rescaled to 0-100. The PACT-Q2 is to be administered to patients once treatment is ongoing. Due to the non-normality of the data, results presented are for median change instead of mean change in PACT-Q2 scores from baseline (V1) to Initiation stage (V2) and from baseline (V1) to Continuation stage (V3) with full range instead of standard deviation of the differences.
Time Frame: From baseline up to 210 days
Population: Main Analysis set (MAS): This includes all eligible patients who met inclusion/exclusion criteria with known assigned treatment information.
Measure: Median (Full Range); unit: Unit on scale
Arm/Group | Cohort A
Number analyzed (Participants) | 4100
Unit on scale
  Median change from V1 to V2: number analyzed (Participants) | 3992
  Median change from V1 to V2 | 19.23 [-67.3 to 86.5]
  Median change from V1 to V3: number analyzed (Participants) | 3827
  Median change from V1 to V3 | 23.08 [-82.7 to 92.3]
Statistical Analysis 1: Comparison: Cohort A; Statistical analysis for median change in PACT-Q2 scores from V1 to V2; Test type: Other; p < 0.0001, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test has been used for this analysis
Statistical Analysis 2: Comparison: Cohort A; Statistical analysis for median change in convenience PACT-Q2 scores from V1 to V3; Test type: Other; p < 0.0001, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test has been used for this analysis

2. Primary Outcome: Satisfaction PACT-Q2 Scores at Second and Last Assessment Compared to Baseline Assessment
Description: as for outcome 1
Time Frame: From baseline up to 210 days
Population: as for outcome 1
Measure: Median (Full Range); unit: Unit on scale
Arm/Group | Cohort A
Number analyzed (Participants) | 4100
Unit on scale
  Median change from V1 to V2: number analyzed (Participants) | 3992
  Median change from V1 to V2 | 17.86 [-85.7 to 78.6]
  Median change from V1 to V3: number analyzed (Participants) | 3827
  Median change from V1 to V3 | 21.43 [-57.1 to 85.7]
Statistical Analysis 1: Comparison: Cohort A; Statistical analysis for median change in satisfaction PACT-Q2 scores from V1 to V2; Test type: Other; p < 0.0001, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test has been used for this analysis
Statistical Analysis 2: Comparison: Cohort A; Statistical analysis for median change in satisfaction PACT-Q2 scores from V1 to V3; Test type: Other; p < 0.0001, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test has been used for this analysis

3. Primary Outcome: Convenience PACT-Q2 Scores at Second and Last Assessment Between Treatment Groups
Description: as for outcome 1
Time Frame: Day 30 up to Day 210
Population: as for outcome 1
Measure: Median (Full Range); unit: Unit on scale
Arm/Group | Cohort B- Pradaxa® | Cohort B- VKA
Number analyzed (Participants) | 3179 | 2186
Unit on scale
  V2: number analyzed (Participants) | 2817 | 2016
  V2 | 82.69 [0.0 to 100.0] | 50.00 [3.8 to 100.0]
  V3: number analyzed (Participants) | 2709 | 1944
  V3 | 86.54 [15.4 to 100.0] | 59.62 [0.0 to 100.0]
Statistical Analysis 1: Comparison: Cohort B- Pradaxa® vs Cohort B- VKA; Mean change in convenience PACT-Q2 scores between VKA and Pradaxa therapy at initiation stage (V2); Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 18.377, Standard Error of Mean 0.514 — The primary analysis of PACT-Q2 scores was based on the random intercept model, where the matched group is considered as a random effect, the treatment as a fixed effect and the score as the response variable
Statistical Analysis 2: Comparison: Cohort B- Pradaxa® vs Cohort B- VKA; Mean change in convenience PACT-Q2 scores between VKA and Pradaxa therapy at continuation stage (V3); Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 23.341, Standard Error of Mean 0.509 — [estimate comment as in outcome 3, analysis 1]

4. Primary Outcome: Satisfaction PACT-Q2 Scores at Second and Last Assessment Between Treatment Groups
Description: as for outcome 1
Time Frame: Day 30 up to Day 210
Population: as for outcome 1
Measure: Median (Full Range); unit: Unit on scale
Arm/Group | Cohort B- Pradaxa® | Cohort B- VKA
Number analyzed (Participants) | 3179 | 2186
Unit on scale
  V2: number analyzed (Participants) | 2817 | 2016
  V2 | 67.86 [0.0 to 100.0] | 50.00 [0.0 to 100.0]
  V3: number analyzed (Participants) | 2709 | 1944
  V3 | 71.43 [17.9 to 100.0] | 50.00 [0.0 to 100.0]
Statistical Analysis 1: Comparison: Cohort B- Pradaxa® vs Cohort B- VKA; Mean change in satisfaction PACT-Q2 scores between VKA and Pradaxa therapy at initiation stage (V2); Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 15.884, Standard Error of Mean 0.388 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Cohort B- Pradaxa® vs Cohort B- VKA; Mean change in satisfaction PACT-Q2 scores between VKA and Pradaxa therapy at continuation stage (V3); Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 19.011, Standard Error of Mean 0.408 — [estimate comment as in outcome 3, analysis 1]

5. Primary Outcome: Characterization of Patients With Respect to Congestive Heart Failure, Hypertension, Age (≥75), Diabetes Mellitus, Stroke/Transient Ischemic Attack (TIA), Vascular Disease, Age 65-75, Sex Category (CHA2DS2-VASc) Score
Description: CHA2DS2-VASc score, are clinical prediction rules for estimating the risk of stroke in patients with non-rheumatic atrial fibrillation (AF), a common and serious heart arrhythmia associated with thromboembolic stroke. Such a score is used to determine whether or not treatment is required with anticoagulation therapy or antiplatelet therapy. CHA2DS2-VASc stroke risk score may range from 0 to 9 with 0 being the best outcome. Score of < 2 was considered as low or intermediate risk and score of ≥ 2 was considered as high risk.
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: Percentage of patients (%)
Arm/Group | Cohort A | Cohort B- Pradaxa® | Cohort B- VKA
Number analyzed (Participants) | 4100 | 3179 | 2186
Percentage of patients (%)
  High risk (Score >= 2) | 88.3 | 87.8 | 91.4
  Low risk (Score < 2) | 5.4 | 8.2 | 7.0
  Data not available | 6.3 | 4.0 | 1.6

6. Primary Outcome: Characterization of Patients With Respect to Hypertension, Abnormal Renal and Liver Function, Stroke, Bleeding History or Predisposition, Labile International Normalized Ratio (INR), Elderly (>65 Years), Drug and Alcohol (HAS-BLED) Score
Description: HAS-BLED is a scoring system developed to assess 1-year risk of major bleeding in patients with atrial fibrillation. A calculated HAS-BLED score is between 0 and 9 and based on eight parameters with a weighted value of 0-2. A high score corresponds to a greater risk, while low score corresponds to a lower risk. Data presented are percentage of patients with high and low risk.
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: Percentage of patients (%)
Arm/Group | Cohort A | Cohort B- Pradaxa® | Cohort B- VKA
Number analyzed (Participants) | 4100 | 3179 | 2186
Percentage of patients (%)
  High risk (Score >= 3) | 59.2 | 29.1 | 31.3
  Low risk (Score < 3) | 31.0 | 64.8 | 65.7
  Data not available | 9.7 | 6.8 | 2.9

7. Primary Outcome: Characterization of Patients With Respect to Kidney Function (Creatinine Clearance)
Description: Creatinine is a waste product produced by muscles from the breakdown of a compound called creatine. Creatinine is filtered from the blood by the kidneys and released into the urine. A creatinine clearance test measures creatinine levels in both a sample of blood and a sample of urine from a 24-hour urine collection. The results are used to calculate the amount of creatinine that has been cleared from the blood and passed into the urine. Data presented here are geometric mean and confidence interval of creatinine clearance for patients at baseline (V1), initiation stage (V2) and continuation stage (V3).
Time Frame: Baseline and up to 210 days
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: millilitre per minute (mL/min)
Groups:
- Cohort B- Pradaxa: Newly diagnosed patients with Non-Valvular Atrial Fibrillation (NVAF) and initiated Pradaxa® 110 mg and Pradaxa® 150 mg hard capsules twice daily containing Dabigatran etexilate (active ingredient: Dabigatran) therapy were included.
- Cohort B-VKA: Newly diagnosed patients with Non-Valvular Atrial Fibrillation (NVAF) and initiated Vitamin K Antagonist (VKA) therapy were included.
Arm/Group | Cohort A | Cohort B- Pradaxa | Cohort B-VKA
Number analyzed (Participants) | 4100 | 3179 | 2186
millilitre per minute (mL/min)
  V1: number analyzed (Participants) | 3501 | 2721 | 1813
  V1 | 73.89 [73.02 to 74.77] | 76.24 [75.25 to 77.24] | 71.83 [70.63 to 73.04]
  V2: number analyzed (Participants) | 1318 | 937 | 603
  V2 | 74.59 [73.17 to 76.05] | 75.27 [73.71 to 76.86] | 71.86 [69.87 to 73.89]
  V3: number analyzed (Participants) | 1539 | 1070 | 686
  V3 | 72.82 [71.61 to 74.05] | 74.24 [72.81 to 75.69] | 71.79 [69.98 to 73.63]

8. Primary Outcome: Characterization of Patients With Respect to Comorbidities
Description: Comorbidity is the presence of one or more additional diseases or disorders co-occurring with (that is, concomitant or concurrent with) a primary disease or disorder. Data presented here are percentage of total patients with comorbidities.
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: Percentage of patients (%)
Arm/Group | Cohort A | Cohort B- Pradaxa® | Cohort B- VKA
Number analyzed (Participants) | 4100 | 3179 | 2186
Percentage of patients (%) | 86.4 | 83.4 | 90.9

9. Primary Outcome: Characterization of Patients With Respect to Concomitant Therapies
Description: Concomitant therapies are two or more drugs used or given at or almost at the same time. The data presented here are percentage of total patients for taking concomitant medication.
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: Percentage of patients (%)
Arm/Group | Cohort A | Cohort B- Pradaxa® | Cohort B- VKA
Number analyzed (Participants) | 4100 | 3179 | 2186
Percentage of patients (%) | 86.4 | 83.4 | 91.2

10. Primary Outcome: Characterization of Patients With Respect to Dosing of Pradaxa
Description: The data presented in this outcome measure is percentage of patients in both cohorts receiving 110 mg and 150 mg dose of Pradaxa at baseline (V1).
Time Frame: Baseline and up to 210 days
Population: as for outcome 1
Measure: Number; unit: Percentage of patients (%)
Groups:
- Cohort B: Newly diagnosed patients with Non-Valvular Atrial Fibrillation (NVAF) and initiated Pradaxa® 110 mg and Pradaxa® 150 mg hard capsules twice daily containing Dabigatran etexilate (active ingredient: Dabigatran) therapy were included.
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 4100 | 3179
Percentage of patients (%)
  Pradaxa 110 mg at V1 | 34.9 | 30.4
  Pradaxa 150 mg at V1 | 65.1 | 69.6

11. Primary Outcome: Duration in Months of Previous VKA Treatment
Description: The data presented in this outcome measure are Mean (SD) of duration in months of previous VKA treatment in total patients in cohort A.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Cohort A
Number analyzed (Participants) | 4100
Months | 34.00 (39.93)

12. Secondary Outcome: PACT-Q2 Scores at Last Assessment Compared to Second Assessment
Description: The individual questions in PACT-Q2 were grouped into two domains, convenience and satisfaction. For each domain, a global score was calculated and used for analysis. The range of the global score is 0-100, with higher score indicating better outcome. The global score is calculated by summing up the individual scores, and then rescaled to 0-100. Due to the non-normality of the data, results presented here are median change in PACT-Q2 scores between initiation stage (V2) and Continuation stage (V3).
Time Frame: From 30 days up to 210 days
Population: as for outcome 1
Measure: Median (Full Range); unit: Unit on scale
Arm/Group | Cohort A
Number analyzed (Participants) | 4100
Unit on scale
  Convenience PACT-Q2: number analyzed (Participants) | 3820
  Convenience PACT-Q2 | 1.92 [-80.8 to 82.7]
  Satisfaction PACT-Q2: number analyzed (Participants) | 3820
  Satisfaction PACT-Q2 | 3.57 [-57.1 to 85.7]
Statistical Analysis 1: Comparison: Cohort A; Median convenience and satisfaction PACT-Q2 scores at last assessment compared to second assessment; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test has been used for this analysis

13. Primary Outcome: Stroke- and/or Bleeding Related Risk Factors in Medical History and at Baseline (Not Applicable)
Description: This endpoint is not assessable as the necessary data was not collected in the database
Time Frame: Baseline
Population: Treated set (Necessary data was not collected in the data base)
Arm/Group | Cohort A | Cohort B- Pradaxa® | Cohort B- VKA
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Description of PACT-Q1 Items at Baseline
Description: Patients in Cohort B were given PACT-Q1 to assess patients' expectation from Anticoagulation therapy. Following are the seven items from PACT-Q1. The score range is 1-5. Each question is analyzed individually, with higher score indicating better outcome. A1 - How confident are you that your anticoagulant treatment (AT) will prevent blood clots? A2 - Do you expect that your AT will relieve some of the symptoms you experience? A3 - Do you expect that your AT will cause side effects such as minor bruises or bleeding? A4 - How important is it for you to have an AT that is easy to take? A5 - How concerned are you about making mistakes when taking your AT? A6 - How important is it for you to take care of your AT by yourself? A7 - How concerned are you about how much you may have to pay for your AT? For questions A1, A2, A4 and A6, higher score is higher expectations of the treatment and for questions A3, A5 and A7, lower score is higher expectations of the treatment.
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: Percentage of patients (%)
Arm/Group | Cohort B- Pradaxa® | Cohort B- VKA
Number analyzed (Participants) | 3179 | 2186
Percentage of patients (%)
  A1- Missing | 2.2 | 2.4
  A1- Not at all | 2.0 | 3.1
  A1- A little | 9.6 | 13.0
  A1- Moderately | 27.8 | 31.9
  A1- A lot | 50.8 | 43.4
  A1- Extremely | 7.7 | 6.1
  A2- Missing | 2.2 | 2.4
  A2- Not at all | 11.6 | 11.8
  A2- A little | 18.5 | 23.4
  A2- Moderately | 28.9 | 31.2
  A2- A lot | 30.9 | 26.6
  A2- Extremely | 7.9 | 4.6
  A3- Missing | 2.2 | 2.4
  A3- Not at all | 17.8 | 13.2
  A3- A little | 38.4 | 38.9
  A3- Moderately | 26.9 | 30.7
  A3- A lot | 12.6 | 12.0
  A3- Extremely | 2.2 | 2.6
  A4- Missing | 2.2 | 2.4
  A4- Not at all | 3.3 | 2.7
  A4- A little | 5.6 | 7.3
  A4- Moderately | 16.4 | 20.5
  A4- A lot | 56.1 | 53.0
  A4- Extremely | 16.5 | 14.1
  A5- Missing | 2.2 | 2.4
  A5- Not at all | 17.3 | 11.3
  A5- A little | 25.3 | 23.0
  A5- Moderately | 19.8 | 27.6
  A5- A lot | 27.2 | 27.5
  A5- Extremely | 8.2 | 8.3
  A6- Missing | 2.2 | 2.4
  A6- Not at all | 3.7 | 3.2
  A6- A little | 7.9 | 7.8
  A6- Moderately | 17.3 | 24.9
  A6- A lot | 52.6 | 49.8
  A6- Extremely | 16.3 | 11.9
  A7- Missing | 2.2 | 2.4
  A7- Not at all | 11.4 | 8.8
  A7- A little | 14.8 | 11.1
  A7- Moderately | 31.0 | 20.9
  A7- A lot | 26.2 | 36.9
  A7- Extremely | 14.4 | 20.0

ADVERSE EVENTS:
Time Frame: From first drug administration, until end of the study, up to 210 days.
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment. The safety analysis set including all the patients with actual follow up were used for this analysis.
Groups:
- Cohort B: Newly diagnosed patients with Non-Valvular Atrial Fibrillation (NVAF) and initiated Pradaxa® 110 mg and Pradaxa® 150 mg hard capsules twice daily containing Dabigatran etexilate (active ingredient: Dabigatran) or Vitamin K Antagonist (VKA) therapy were included.
Arm/Group | Cohort A | Cohort B- Pradaxa® | Cohort B- VKA | Cohort B
All-Cause Mortality (participants affected / at risk) | 5/4066 | 2/3164 | 4/2181 | 6/5345
Serious Adverse Events (participants affected / at risk) | 26/4066 | 25/3164 | 15/2181 | 40/5345
Other Adverse Events (participants affected / at risk) | 0/4066 | 0/3164 | 0/2181 | 0/5345
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=4066) | Cohort B- Pradaxa® (N=3164) | Cohort B- VKA (N=2181) | Cohort B (N=5345)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 2 | 3
Atrioventricular block (Cardiac disorders) | 1 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 3 | 2 | 1 | 3
Myocarditis (Cardiac disorders) | 0 | 1 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 2 | 2 | 4
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 1 | 1
Chest discomfort (General disorders) | 0 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 1 | 1 | 2
Death (General disorders) | 1 | 2 | 3 | 5
Sudden death (General disorders) | 1 | 0 | 0 | 0
Appendiceal abscess (Infections and infestations) | 0 | 1 | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pseudomembranous colitis (Infections and infestations) | 0 | 1 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Arteriogram coronary (Investigations) | 0 | 1 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 1
Cerebrovascular disorder (Nervous system disorders) | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 1 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 3 | 4 | 1 | 5
Transient ischaemic attack (Nervous system disorders) | 0 | 2 | 0 | 2
Calculus bladder (Renal and urinary disorders) | 0 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 | 0 | 0 | 0
Cardioversion (Surgical and medical procedures) | 0 | 1 | 0 | 1
Left atrial appendage occlusion (Surgical and medical procedures) | 0 | 1 | 0 | 1
Meningioma surgery (Surgical and medical procedures) | 1 | 0 | 0 | 0
Transurethral prostatectomy (Surgical and medical procedures) | 0 | 1 | 0 | 1
Vascular stent insertion (Surgical and medical procedures) | 1 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
Improper dose reduction in patients not fulfilling reduction criteria, Selection bias, Missing data, Creatinine clearance in minimals, Antiarrhythmic medication contraindicated to Pradaxa, Unassessable Stroke/bleeding related risk factors endpoint

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT02684981/SAP_000.pdf
  • Study Protocol (2015-07-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT02684981/Prot_001.pdf